CLINICAL TRIAL: NCT03169387
Title: Body Composition of Individuals With Cardiovascular Diseases Submitted to Conventional Cardiac or Virtual Reality Rehabilitation: A Randomized Clinical Trial
Brief Title: Body Composition of Individuals With Cardiovascular Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Oeste Paulista (Other)
Responsible Party: Principal Investigator, Ana Paula Coelho Figueira Freire, Professor, Universidade do Oeste Paulista
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35632017
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Diseases; Body Composition
Keywords: Virtual Reality Exposure Therapy
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Microsoft's Xbox 360® will be used with Kinect™,
  Interventions: Behavioral: Virtual Reality
- Conventional Training (Active Comparator): treadmills (embreex) will be used to perform the aerobic training for a period of 30 minutes and free weights and weight training equipment for the resistance training
  Interventions: Behavioral: Conventional Training

INTERVENTIONS:
Behavioral: Virtual Reality — For the VRG training, Microsoft's Xbox 360® will be used with Kinect™, which features an infrared camera sensor that recognizes user movements without a controller. The games used will be YourShape™(Fitness Evolved) and Dance Central 3™, which will be played for 25 minutes each; the former will be associated with the use of Velcro weights on the ankles and dumbbells in the hands to provide resistance.
  Other Names: Experimental: Virtual Reality
  Arms: Virtual Reality
Behavioral: Conventional Training — treadmills (embreex) will be used to perform the aerobic training for a period of 30 minutes and free weights and weight training equipment for the resistance training, which will be carried out in 3 sets of 10 repetitions, with a recovery interval of 1 minute between sets.
  Other Names: Active Comparator: Conventional Training
  Arms: Conventional Training

SUMMARY:
Introduction: Cardiovascular diseases are the leading cause of death in the world, thus, rehabilitation programs are essential to improve symptoms and reduce mortality. Virtual reality presents itself as a new alternative of therapeutic resource, stimulating the practice of physical activity through interaction between man and machine, based on the use of games and virtual environments. Objective: To compare the body composition of individuals with cardiovascular diseases submitted to conventional cardiac or virtual reality rehabilitation. Methods: Twenty-four individuals with cardiovascular diseases, divided into a conventional rehabilitation group (GRC) or virtual reality rehabilitation group (GRV), will be evaluated, and undergo a rehabilitation program for a period of 8 weeks, with two weekly sessions lasting 60 minutes. For the GRV training, the Xbox 360® from Microsoft with Kinect™ will be used with the games YourShape™ (Fitness Evolved) and Dance Central 3™. For the GRC training, treadmills (embreex) will be used to perform the aerobic training and free weights and weight training equipment to perform the resistance training. Food frequency will be evaluated by means of the Food Frequency Questionnaire, food consumption by the 24-hour food recall, body composition by bioimpedance, and functional capacity by the six-minute walk test. For analysis of data normality the Shapiro Wilk test will be applied. For paired analysis, the Student's T test will be performed in case of normal distribution or the Wilcoxon test for variables that do not follow Gaussian distribution. The intergroup comparisons will be analyzed through absolute variation before and after the interventions and the unpaired Student's T test or Mann Whitney test applied according to the normality of the data. The level of significance adopted will be 5%.

DETAILED DESCRIPTION:
Materials and methods Ethical aspects Participants included in the study will be instructed in relation to all procedures that will be performed and sign the informed consent form agreeing to participate in the study (Annex 1), which was approved by the Institutional Ethics Committee (CAAE: CAAE 62437816.4.0000.5515,protocol number 1.865.530) and is in line with CONEP resolution 466/2012.

Experimental design In the first instance, the patients will perform an initial evaluation (Appendix 2) for the detection of comorbidities, diagnosis identification, clinical history, and collection of drug data. The following will be evaluated before and after 8 weeks of intervention: food frequency, food consumption, anthropometric variables, abdominal circumference, body composition, glycemic behavior, and functional capacity.

Food frequency The Food Frequency Questionnaire (FFQ) will be used to analyze the periodicity of food consumption. The FFQ has a space that contains the food and another for the respondent to register how often they consume this food. The frequency is recorded in units of time: days, weeks, months, years, according to the needs of the evaluation. It is considered a practical and easily applied questionnaire, besides being important for studies that associate diet with chronic diseases .

Food consumption The 24-hour food recall (R24h) will be used to measure the current food consumption of the individuals. The R24h is a quantitative assessment of food and beverage intake. It provides detailed information on weight and total volume of portions consumed in the previous 24 hours. This method aims to evaluate the current diet and estimate absolute or relative values of nutrient intake, according to the total of the foods offered to the individual. The recall will be completed by the patients for three consecutive days.

Anthropometric variables Weight and height will be evaluated through anthropometry, using a Filizola® scale (accuracy of 100g), with the patient wearing light, comfortable clothes and barefoot. Height will be measured using a Filizola® stadiometer (0.1 cm accuracy) with the patient barefoot, in the orthostatic position, their back to the marker, feet together, head adjusted to the Frankfurt plane, and the metal bar on the patient's head. The body mass index (BMI) will be calculated based on the patient's weight and height, through the weight / height ratio.

Abdominal circumference The abdominal circumference will be obtained using a non-distensible tape measure (accuracy of 1 mm). With the individual in the orthostatic position, feet parallel, upper limbs relaxed and alongside the trunk, the tape measure will be positioned at the height of the iliac crest and immediately above the umbilical scar, without compressing the skin. The measurement will be performed 3 times and the lowest value selected for the study.

Body composition Body composition will be evaluated using Tetrapolar Bioimpedance Apparatus (BIA), Biodynamics® Model 310e, in which weight and percentage of body fat and fat free weight (muscles, bones, and organs) will be analyzed and quantified. The BIA will be performed in the morning and patients will be required to be in a fasting state, empty their bladder prior to the test, discontinue diuretic medication 24 hours prior to the test, refrain from drinking alcohol and caffeine for 24 hours prior to the examination, and not perform intense physical activity for 72 hours before the evaluation. The BIA will not be performed on patients with pacemakers or those with unstable heart failure, as alterations in volume could interfere with the results.

Glycemic behavior Verification of capillary glycemia will be carried out using a glycosimeter, brand OptiumXceed®, that determines glucose in fresh capillary blood, collected by puncturing the digital pulp of the ring finger using sterile lancet blades. The collections will be carried out individually, before and after the training.

Functional capacity Functional capacity will be evaluated through the 6-minute Walk Test (WT6') performed according to the criteria established by the American Thoracic Society. The WT6' will be performed in a hall of the gymnasium at the Universidade do Oeste Paulista, Presidente Prudente/SP- Brazil.

Cardiovascular parameters Heart rate will be measured using a Sigma® heart rate monitor. Oxygen saturation will be verified through a Choicemmed® brand pulse oximeter, model Md300c1. Blood pressure will be checked with the patient seated, in the dominant arm, using a Premium® brand aneroid sphygmomanometer and Littman® brand stethoscope, according to the Brazilian arterial hypertension guidelines.

Training protocol For both groups the training protocol will consist of 2 weekly sessions, lasting 60 minutes, for a period of 8 weeks in the Physical Therapy Clinic of the Universidade do Oeste Paulista, Presidente Prudente/SP, Brazil, totaling sixteen sessions. The initial and final 5 minutes of each session will be used to measure blood pressure, blood glucose, and O2 saturation, and apply the Borg scale of subjective effort. Throughout all sessions, the Borg scale of subjective effort and heart rate will also be verified to ensure that the training heart rate, calculated individually according to the Karvonen formula, is not exceeded.

For the GVR training, Microsoft's Xbox 360® will be used with Kinect™, which features an infrared camera sensor that recognizes user movements without a controller. The games used will be YourShape™(Fitness Evolved) and Dance Central 3™, which will be played for 25 minutes each; the former will be associated with the use of Velcro weights on the ankles and dumbbells in the hands to provide resistance.

For the GRC training, treadmills (embreex) will be used to perform the aerobic training for a period of 30 minutes and free weights and weight training equipment for the resistance training, which will be carried out in 3 sets of 10 repetitions, with a recovery interval of 1 minute between sets. The exercises performed will be shoulder abduction, elbow flexion, and knee extension and flexion, all performed in the seated position, with the exception of the knee flexion which will be performed in the orthostatic position. The increase in resistance will be carried out in an individualized way based on the Borg sensation of effort (13- slightly tiring).

Statistical analysis The data will be analyzed using the statistical software GraphPadPrism. For analysis of data normality the Shapiro Wilk test will be applied. For paired analysis, the Student's T test will be performed in case of normal distribution or the Wilcoxon's test for variables that do not follow Gaussian distribution. The intergroup comparisons will be analyzed by absolute variation before and after the interventions and the unpaired Student's T test or Mann Whitney test applied according to normality of the data. The level of significance used will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 45 years of age,
* Both genders,
* Presenting cardiovascular diseases (coronary insufficiency, postoperative myocardial revascularization, acute myocardial infarction, systemic arterial hypertension, and diabetes mellitus)
* Patients hemodynamically stable,
* Not participated in previous rehabilitation programs for the last year,
* Not present arteriopathies or muscular or orthopedic alterations.

Exclusion Criteria:

* Decompensation during the training protocol,
* Patients who do not adapt to the training,
* Patients a participation frequency of less than 75%

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in percentual of body fat | Baseline and 8 weeks of training
  Body composition

SECONDARY OUTCOMES:
Change in fat free weight | Baseline and 8 weeks of training
  Body composition

OTHER OUTCOMES:
Change in abdominal circumference | Baseline and 8 weeks of training
  Mesurement of abdmominal region

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Paula Coelho Figueira Freire, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plans for sharing data with other reserarchers